CLINICAL TRIAL: NCT06921239
Title: HLA Antibodies in Systemic Lupus Erythematosus
Acronym: LEDHLA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0043
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: HLA Antibodies; Systemic Lupus Erythematosus
Keywords: HLA antibodies; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients suffering from autoimmune diseases show false-positive results when anti-HLA antibodies are identified. This false positivity makes it difficult to obtain an organ transplant based on immunological compatibility (absence of anti-HLA antibodies directed against graft antigens). The objectives of this project are to study the prevalence of these false positivities in a population of lupus patients, and to evaluate biological tests that can negate these false positivities.

ELIGIBILITY:
Inclusion Criteria:

* Patients Adults
* Followed in the internal medicine department of Amiens University Hospital - With systemic lupus erythematosus
* Without HLA immunization risk factors (no history of pregnancy, transfusions or transplants)
* With sera stored in the biobank

Exclusion Criteria:

* minor Patients
* Opposing the re-use of their personal data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Adults - Followed in the internal medicine department of Amiens University Hospital - With systemic lupus erythematosus - Without HLA immunization risk factors (no history of pregnancy, transfusions or transplants) - With sera stored in the biobank
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
prevalence of unexplained antibody positivity | 6 months
  prevalence of unexplained antibody positivity

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No